CLINICAL TRIAL: NCT04565171
Title: A Single-center, Non-randomized, Open-Label, Single-Dose Study to Evaluate the Pharmacokinetics of Yimitasvir Phosphate Capsule in Subjects With Normal Renal Function and End-stage Renal Disease Without Hemodialysis
Brief Title: Pharmacokinetics of Yimitasvir Phosphate Capsule in Subjects With Normal Renal Function and ESRD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCD-DDAG181PA-18-001
Record Dates: First submitted 2020-09-22; First posted 2020-09-25 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2020-09

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — yimitasvir

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants with renal impairment (Experimental): Participants with End-stage renal disease will receive a single dose of Yimitasvir Phosphate Capsule.
  Interventions: Drug: Yimitasvir Phosphate Capsule
- Participants with normal renal function (Experimental): Participants with normal renal function will receive a single dose of Yimitasvir Phosphate Capsule.
  Interventions: Drug: Yimitasvir Phosphate Capsule

INTERVENTIONS:
Drug: Yimitasvir Phosphate Capsule — DAG181 100 mg (100 mg Capsule) administered orally
  Other Names: DAG181

SUMMARY:
This study is to evaluate the single-dose pharmacokinetics (PK) and safety of Yimitasvir phosphate capsule in participants with End-stage renal disease without hemodialysis using matched healthy participants as a control group.

ELIGIBILITY:
Inclusion Criteria:

1. male or female, age 18 to 70 years of age, inclusive;
2. must have a calculated body mass index (BMI) from 18 to 28 kg/m2 at study screening;
3. Glomerular filtration rate must be < 15 mL/min /1.73 m2 for End-stage renal disease without hemodialysis group, and ≥ 90 mL/min for Normal Renal Function group(using MDRD method);
4. matched for age (±5 years) ,gender and BMI(±15%) with a subject in the End-stage renal disease without hemodialysis group;

Exclusion Criteria:

1. allergies constitution ( multiple drug and food allergies);
2. Use of >5 cigarettes per day during the past 3 months;
3. A positive test results for HbsAg, Hepatitis C antibody, HIV-1 antibody, or Treponema pallidum antibody；
4. History of alcohol abuse；
5. Donation or loss of blood over 400 mL within 3 months prior to the first dose of study drug；
6. Subjects deemed unsuitable by the investigator for any other reason.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2022-05-07 (Actual); Study Completion 2022-05-07 (Actual)

PRIMARY OUTCOMES:
Plasma pharmacokinetics (PK) parameters of DAG181 as measured by AUC | From Days 1-5
  AUC is defined as the concentration of drug area under the curve
Plasma pharmacokinetics (PK) parameters of DAG181 as measured by Cmax | From Days 1-5
  Cmax is defined as the maximum concentration of drug

SECONDARY OUTCOMES:
Incidence of adverse events | From Days 1-5
  The incidence of adverse events will be summarized

CONTACTS AND LOCATIONS:
Overall Officials: jia Miao, Doctor, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No